CLINICAL TRIAL: NCT03497195
Title: Achieving TB Control In Zambia Through Scale Up Of Innovative Tools And Proven Active TB Case Finding Interventions
Brief Title: Achieving Tuberculosis (TB) Control In Zambia
Acronym: TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stewart Reid, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300001132
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community level screening; Arm 1 (Active Comparator): use of chest X-ray plus Xpert Ultra for community level TB screening
  Interventions: Diagnostic Test: Screening at community level
- Community level screening: Arm 2 (Active Comparator): use of C-reactive Protein and Xpert Ultra for community level TB screening
  Interventions: Diagnostic Test: Screening at community level

INTERVENTIONS:
Diagnostic Test: Screening at community level — comparison of chest x-ray and Xpert Ultra versus CRP and Xpert Ultra for active community based screening

SUMMARY:
To achieve TB control, innovative case finding interventions are needed that will reach the broader affected population including those that do not access the health facilities. Systematic community case finding with highly sensitive screening and diagnostic tools are needed. At the facility level, the index of suspicion for TB by health care workers needs to be raised to ensure that all those that need TB screening are appropriately screened.

DETAILED DESCRIPTION:
The purpose of this study is to initiate sustained, active health facility and community-based case finding interventions to achieve improved TB case detection in high burden settings (Zambia) and contribute to TB control.

The interventions are expected to increase the impact of Xpert on TB case finding, thus increase TB case detection through scaling up of a combination of community level and facility level TB case finding interventions. The study will generate evidence on the added value of using Chest X-ray (CXR) screening at community level, whilst also comparing the performance of CXR with computer assisted diagnosis (CAD) and C-reactive protein (CRP) and symptoms as screening tools in terms sensitivity, specificity and cost effectiveness. Symptom screen alone has been shown to be suboptimal for screening as it misses a significant percentage of TB due to atypical presentation of TB in HIV-infected populations.

ELIGIBILITY:
Inclusion Criteria:

-

Program Implementation:

Inclusion criteria:

* Any adult or child with TB symptoms (weight loss, chest pain, shortness of breath, fever, cough, hemoptysis, night sweats)
* Ability to produce sputum
* Verbal consent of parent or guardian if < 18 years old

Operations Research:

Inclusion criteria

* Adults (18 years and older)
* TB symptoms (weight loss, chest pain, shortness of breath, fever, cough, hemoptysis, night sweats)
* Ability to provide a sputum sample
* Willing to provide written informed consent
* Willing to undergo full clinical evaluation
* Willing to undergo a CXR

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18194 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
increase TB case detection | 6 months
  comparison of two diagnostic tools (Chest Xray with CAD versus CRP) and Xpert Ultra for active community based TB case detection

CONTACTS AND LOCATIONS:
Overall Officials: Monde Muyoyeta, MD,PhD, Principal Investigator — Center for Infectious Disease Research in Zambia
Locations (1):
- Center for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229